CLINICAL TRIAL: NCT01976819
Title: Phase 2 Clinical Feasibility Study of a New Speaking Valve With a Heat- and Moisture Exchanger (TW) for Tracheotomized Patients.
Brief Title: Clinical Assessment of New Speaking Valve With Heat and Moisture Exchanger (HME) for Tracheotomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UD788_TW
Record Dates: First submitted 2013-10-17; First posted 2013-11-06 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Tracheostomy
Keywords: Tracheotomy; Tracheostomy; Speaking valve; HME; patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TW speaking valve/HME (Experimental): Use of the TW speaking valve/HME
  Interventions: Device: TW speaking valve/HME

INTERVENTIONS:
Device: TW speaking valve/HME — The TW speaking valve with HME will be used during the day, whereas during sleep patients will use an HME without an automatic speaking valve. Data from TW15 and TW22 will be combined.
  Other Names: DualCare speaking valve/HME

SUMMARY:
This clinical investigation addresses the performance of a re-designed The current study aims to investigate the next version of the TW speaking valve, in combination with both a 15mm and 22mm HME cassette.

DETAILED DESCRIPTION:
This clinical investigation addresses the performance of a re-designed (updated) speaking valve with Heat and Moisture Exchangers (HME) for tracheotomized patients (project development name 'TW', commercial name 'DualCare'). Study participants trial the new device for 2 weeks after which they can choose to discontinue using the device or continue in the 3 month follow-up part of the study. Clinical feasibility is assessed using structured questionnaires addressing voice and speech, quality of life, breathing, swallowing, olfaction, sleeping, and respiratory symptoms. This is an exploratory, observational study and no specific hypotheses have been formulated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* has a tracheostomy
* is spontaneously breathing
* has a cuffless tracheostomy tube
* has a tracheostomy tube with inner and outer cannula
* currently uses an HME and/or speaking valve

Exclusion Criteria:

* patient unable to handle or remove the device him/herself when needed, e.g. has decreased level of cognition or reduced mobility of the arms and/or hands
* is mechanically ventilated in any way
* has a tidal volume of less than 100 ml
* is suffering from severe aspiration
* is laryngectomized: the device will block the possibility to exhale if speaking mode is unintentionally activated
* has severe upper airway obstruction, this may cause air trapping
* has thick and copious secretions which might block the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardus FA van der Laan, PhD, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymous (de-identified) patient data will be used for publication, expected 2016.

RESULTS

PARTICIPANT FLOW:
Groups:
- TW Speaking Valve/HME: At baseline, participants were asked to complete a baseline questionnaire. After that, patients were asked to use both the current (old) TW15 or the TW22 for a week. After each week, patients completed a device specific questionnaire. At the end of the two week period, patients also completed a structured and comparative questionnaire.
  Patients were then asked to use the new updated Speaking Valve for a week and then to complete relevant sections of the same questionnaire that was also used for the previous (old) device. Patients could decide again whether they wanted to participate in the long term part of the study, which will follow the same structure with the same questionnaires as in Stage 0.
Period: Overall Study
Arm/Group | TW Speaking Valve/HME
Started | 16
Completed | 11
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- TW Speaking Valve/HME: Use of the TW speaking valve/HME
  TW speaking valve/HME: The TW speaking valve with HME will be used during the day, whereas during sleep patients will use an HME without an automatic speaking valve
Arm/Group | TW Speaking Valve/HME
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.50 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Region of Enrollment [Number; unit: participants]
  Netherlands | 16

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Patient Experiences Associated With Exposure to the Speaking Valve With a Heat- and Moisture Exchanger (TW) for Tracheotomized Patients Based on Results From Questionnaires.
Description: Patients were asked to use either the old TW15 and the TW22 HME device for a week, data combined for the two devices (the device used was recorded). After each week, patients completed a device specific questionnaire (Borg Scale).
  After the re-design (ie Updated speaking valve), patients were asked to use the new Speaking Valve for a week and then to complete relevant sections of the same questionnaire. Both at baseline and in the follow-up, patients were asked about their breathing using a Borg scale at a particular moment. This scale has a range from 0-6 where a score close to "0" indicates less breathing problems.
Time Frame: 3 weeks including Baseline, week 1, 2 (old device) and week 3 (updated device).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Updated Speaking Valve/HME: Use of the updated speaking valve/HME
  TW speaking valve/HME: The TW speaking valve with HME will be used during the day, whereas during sleep patients will use an HME without an automatic speaking valve. Data from TW15 and 22 combined.
- Use of the Old HME Speaking Valve: Data from the use of the old HME speaking valve, data from TW15 and TW22 combined.
Arm/Group | Updated Speaking Valve/HME | Use of the Old HME Speaking Valve
Number analyzed (Participants) | 11 | 16
units on a scale
  Breathing with TW follow-up | 0.5 (0.8) | 1.1 (0.5)
  Breathing with TW baseline | 2.3 (1.9) | 2.3 (1.9)

2. Primary Outcome: Hours of HME Use Per Day.
Description: The mean number of hours of TW use per 24 hours was calculated.
Time Frame: Weeks 1 and 2 (Old device, data averaged) and Week 3 (Updated device)
Measure: Mean (Standard Deviation); unit: hours per day
Groups:
- Use of Updated Speaking Valve: Use of the TW speaking valve/HME
  TW speaking valve/HME: The TW speaking valve with HME will be used during the day, whereas during sleep patients will use an HME without an automatic speaking valve. Data from TW15 and 22 combined.
- Use of Old Speaking Valve: Usage of the old speaking valve device. TW15 and TW22 combined.
Arm/Group | Use of Updated Speaking Valve | Use of Old Speaking Valve
Number analyzed (Participants) | 11 | 16
hours per day | 13.5 (2.7) | 14.1 (2.3)

3. Primary Outcome: Device Preference Rating.
Description: Patients were asked to rate the devices on a scale from 0-10, where "10" indicates the best score and "0" the worst score. The overall mean satisfaction with the speaking valve was rated.
Time Frame: Weeks 1 and 2 (Old device, data averaged) and Week 3 (Updated device)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Use of Updated Speaking Valve: Use of the TW speaking valve/HME
  TW speaking valve/HME: The TW speaking valve with HME will be used during the day, whereas during sleep patients will use an HME without an automatic speaking valve. Data from TW15 and 22 are combined.
- Use of Old Speaking Valve: Data from TW15 and 22 combined.
Arm/Group | Use of Updated Speaking Valve | Use of Old Speaking Valve
Number analyzed (Participants) | 11 | 16
units on a scale | 8.4 (1.5) | 6.5 (2.5)

ADVERSE EVENTS:
Arm/Group | TW Speaking Valve/HME
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TW Speaking Valve/HME (N=16)
stoma irritation (Skin and subcutaneous tissue disorders) | 1 (1) — stoma irritation occurred when twisting device
sound leakage past cannula (Surgical and medical procedures) | 1 (1) — sound leakage past cannula when coughing

LIMITATIONS AND CAVEATS:
small sample size;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No